CLINICAL TRIAL: NCT05785897
Title: ST-segment Elevation Myocardial infArction Treated With a Polymer-free Sirolimus-based nanocarrieR Eluting Stent and a P2Y12 Inhibitor-based Aspirin-free Single Antiplatelet Strategy Versus Conventional Dual AntiPlatelet Therapy
Brief Title: STEMI Treated With a Polymer-free Sirolimus-coated Stent and P2Y12 Inhibitor-based SAPT Versus Conventional DAPT
Acronym: STARS DAPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IGLESIAS Juan Fernando (Other)
Collaborators: Clinical Trials Unit University of Bern (Unknown)
Responsible Party: Sponsor-Investigator, IGLESIAS Juan Fernando, Principal investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0309
Record Dates: First submitted 2023-03-11; First posted 2023-03-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Single antiplatelet therapy; P2Y12 receptor inhibitor; ST-segment elevation myocardial infarction; Polymer-free drug-eluting stent
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Potent P2Y12 receptor inhibitor-based single antiplatelet therapy (SAPT) (Experimental): * P2Y12 receptor inhibitor-based SAPT with ticagrelor (90 mg bd) or prasugrel (10 mg od, or 5 mg in patients ≥75 years or with a body weight <60 kg), at the discretion of the investigator, during 12 months after the index procedure.
  * Clopidogrel-based SAPT will not be allowed.
  * Aspirin will be discontinued after primary PCI, or at latest at hospital discharge.
  Interventions: Device: Successful primary PCI, defined as primary PCI of the culprit lesion with ≥1 Abluminus NP polymer-free sirolimus-based nanocarrier eluting stent (Concept Medical Inc., India) implantation
- Conventional dual antiplatelet therapy (DAPT) (Active Comparator): * DAPT combining aspirin (≥75 mg od) and a potent P2Y12 receptor inhibitor, either ticagrelor (90 mg bd) or prasugrel (10 mg od, or 5 mg in patients ≥75 years or with a body weight <60 kg), at the discretion of the investigator, during 6 or 12 months after the index procedure, followed by aspirin-based SAPT.
  * Clopidogrel (75 mg od orally) will be allowed if ticagrelor or prasugrel are contra-indicated or not available.
  Interventions: Device: Successful primary PCI, defined as primary PCI of the culprit lesion with ≥1 Abluminus NP polymer-free sirolimus-based nanocarrier eluting stent (Concept Medical Inc., India) implantation

INTERVENTIONS:
Device: Successful primary PCI, defined as primary PCI of the culprit lesion with ≥1 Abluminus NP polymer-free sirolimus-based nanocarrier eluting stent (Concept Medical Inc., India) implantation — 'All-comer' subjects with acute STEMI undergoing primary PCI according to current ESC guidelines will be eligible.
  Eligible subjects will be pre-treated with DAPT consisting of aspirin (loading dose: 150-300 mg orally or 80-500 mg intravenously, maintenance dose: 75-100 mg daily orally) and a potent P2Y12 receptor inhibitor, either ticagrelor (loading dose: 180 mg orally, maintenance dose: 90 mg bd orally) or prasugrel (loading dose: 60 mg orally, maintenance dose: 10 mg od orally or 5 mg od orally if age >75 years or weight <60 kg) at the time of STEMI diagnosis, or at the very latest at the time of primary PCI.
  Successful primary PCI, defined as primary PCI of the culprit lesion with ≥1 Abluminus NP polymer-free sirolimus-based nanocarrier eluting stent (Concept Medical Inc., India) implantation and final residual stenosis <30% by visual estimation or 20% by QCA.
  Other Names: 'All-comer' subjects with acute STEMI undergoing primary PCI according to current ESC guidelines will be eligible.; Pre-treatment with DAPT consisting of aspirin and a potent P2Y12 receptor inhibitor, either Ticagrelor or Prasugrel at the time of STEMI diagnosis, or at the very latest at the time of primary PCI

SUMMARY:
Primary percutaneous coronary intervention (PCI) is the preferred revascularization strategy for patients with acute ST-segment elevation myocardial infarction (STEMI). Compared with bare-metal stents (BMS) and early-generation thick-strut polymer-based drug-eluting stents (DES), newer-generation DES with thinner strut stent platforms and durable or biodegradable polymers have been shown to improve long-term safety and efficacy outcomes among patients with STEMI. Accordingly, the use of newer-generation DES over BMS is currently recommended by the most recent guidelines. Vessel healing at the culprit site after DES implantation is however substantially delayed in patients with acute STEMI as compared to those with chronic coronary syndromes and is associated with a long-term risk for recurrent stent-related adverse clinical outcomes. These findings highlight the need for future iterations in modern DES technology to further improve clinical outcomes following PCI in this highest-risk patient subset.

Current guidelines recommend dual antiplatelet therapy (DAPT) consisting of aspirin and a potent P2Y12 receptor inhibitor for 12 months after primary PCI for STEMI, unless there are contraindications such as excessive risk of bleeding. A recent meta-analysis of five large-scale randomized clinical trials including a total of 32'145 patients, of whom 4,070 (12.7%) patients were treated for STEMI, indicated that 1-3 months of DAPT followed by P2Y12 inhibitor-based single antiplatelet therapy (SAPT) after second-generation DES implantation in patients with chronic and acute coronary syndromes was associated with lower risk for major bleeding and similar risk for stent thrombosis, all-cause death, myocardial infarction, and stroke compared with conventional DAPT. These findings suggest that a potent P2Y12 inhibitor-based SAPT following a short DAPT course (1-3 months) may represent a preferable treatment option, which is associated with similar ischemic, but lower bleeding risk, for patients undergoing PCI with newer-generation DES compared to standard conventional 12 months DAPT.

The question of whether SAPT using a potent oral P2Y12 inhibitor (ticagrelor or prasugrel) without aspirin (aspirin-free strategy) after primary PCI with a newest-generation thin-strut polymer-free drug-eluting stent is safe and effective compared to a conventional guideline-recommended 6- to 12-month DAPT course among patients with STEMI remains uncertain.

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention (PCI) is the preferred revascularization strategy for patients with acute ST-segment elevation myocardial infarction (STEMI). Compared with bare-metal stents (BMS) and early-generation thick-strut polymer-based drug-eluting stents (DES), newer-generation DES with thinner strut stent platforms and durable or biodegradable polymers have been shown to improve long-term safety and efficacy outcomes among patients with STEMI. Accordingly, the use of newer-generation DES over BMS (class of recommendation I, level of evidence A) is currently recommended by the most recent guidelines of the European Society of Cardiology (ESC) for the management of STEMI. Vessel healing at the culprit site after DES implantation is however substantially delayed in patients with acute STEMI as compared to those with chronic coronary syndromes and is associated with a long-term risk for recurrent stent-related adverse clinical outcomes. These findings highlight the need for future iterations in modern DES technology to further improve clinical outcomes following PCI in this highest-risk patient subset.

Newest-generation DES combining ultrathin-strut cobalt chromium metallic stent platforms with biodegradable polymers were introduced to mitigate chronic inflammation and arterial injury, promote rapid endothelization and improve clinical outcomes following PCI compared with contemporary second-generation durable polymer DES. These features might be particularly important in the enhanced thrombotic and inflammatory environment of acute STEMI and translate into differential clinical outcomes between different DES technologies. In the BIOSTEMI randomized trial, newer-generation biodegradable polymer sirolimus-eluting stents (BP-SES) (Orsiro, Biotronik AG, Switzerland) were found superior to second-generation durable polymer everolimus-eluting stents (DP-EES) (Xience Prime/Expedition, Abbott Vascular, USA) with respect to target lesion failure (TLF) at 1- and 2-year of follow-up among 1,300 patients with acute STEMI undergoing primary PCI, a difference caused by a lower risk for clinically indicated target lesion revascularization. Newest-generation thin-strut polymer-free DES have potential to further mitigate chronic inflammation, promote faster re-endothelialization and reduce DAPT duration, and might represent the future standard-of-care for patients with STEMI undergoing primary PCI. Abluminus DES+ (Concept Medical Inc., India), a novel thin-strut biodegradable polymer sirolimus-eluting stent with a unique Envisolution technology aimed at facilitating early vascular healing. In the en-ABL e-REGISTRY, a large-scale all-comers post-market registry including 2,500 patients, the Abluminus DES+ (Concept Medical Inc., India) showed very low TLF rates (2.2%) among patients with acute myocardial infarction (n=999), suggesting a potential benefit of this newest DES technology in the highest-group of patients with acute coronary syndrome (ACS) with delayed vascular healing. The Abluminus NP (Concept Medical Inc., India) is a novel thin-strut cobalt chromium sirolimus-based nano carrier eluting stent system specially designed to reduce polymer-related inflammation and accelerate vascular healing. In the NANOACTIVE first-in-man study (data not published), the Abluminus NP (Concept Medical Inc., India) has shown promising very low rates of major adverse clinical events among 86 all-comer patients undergoing PCI. However, no dedicated randomized clinical trial to date has evaluated the safety and efficacy of newest-generation thin-strut cobalt chromium polymer-free drug-coated stents for primary PCI in patients with acute STEMI.

2017 ESC guidelines on the management of STEMI recommend dual antiplatelet therapy (DAPT) consisting of aspirin and a potent P2Y12 receptor inhibitor, ticagrelor or prasugrel (or clopidogrel, if ticagrelor or prasugrel are not available or are contraindicated) for 12 months after primary PCI for STEMI, unless there are contraindications such as excessive risk of bleeding (class of recommendation I, level of evidence A). In patients who are at high risk of severe bleeding complications, discontinuation of P2Y12 inhibitor therapy after 6 months may be considered (class of recommendation IIa, level of evidence B). Several randomized clinical trials have investigated alternative antiplatelet therapy strategies for patients with acute STEMI who undergo primary PCI with newer-generation DES. In the DAPT-STEMI randomized, controlled trial, 1,100 STEMI patients who underwent primary PCI with a second-generation DES (Resolute Integrity, Medtronic, USA), and who were event-free at six months on DAPT, were randomized in a 1:1 ratio to aspirin-based single antiplatelet therapy (SAPT) or DAPT for an additional six months. At 18 months, the primary endpoint, a composite of all-cause death, any myocardial infarction, any revascularization, stroke, or Thrombolysis in Myocardial Infarction (TIMI) major bleeding, occurred in 4.8% of patients receiving SAPT and 6.6% of patients receiving DAPT (HR, 0.73; 95% confidence interval (CI), 0.41 to 1.27; p=0.26), meeting the pre-specified study definition for non-inferiority (p for non-inferiority=0.004). In summary, the DAPT-STEMI trial demonstrated that a 6-month DAPT course was non-inferior to standard DAPT for 12 months in patients with event-free STEMI after primary PCI with second-generation DES. However, whether further iterations of DES technology, including thinner-strut stent platforms and biodegradable polymer coatings, may facilitate a shorter DAPT duration with respect of safety (bleeding) and efficacy (ischemic) outcomes has remained uncertain.

A recent meta-analysis of five large-scale randomized clinical trials including a total of 32'145 patients, of whom 4,070 (12.7%) patients were treated for STEMI, indicated that 1-3 months of DAPT followed by P2Y12 inhibitor-based single antiplatelet therapy (SAPT) after second-generation DES implantation in patients with chronic and acute coronary syndromes was associated with lower risk for major bleeding (random-effects model: HR, 0.63; 95%CI, 0.45-0.86) and similar risk for stent thrombosis (random-effects model: HR, 1.19; 95%CI, 0.86-1.65), all-cause death (random-effects model: HR, 0.85; 95%CI, 0.70-1.03), myocardial infarction (random-effects model: HR, 1.05; 95%CI, 0.89-1.23), and stroke (random-effects model: HR, 1.08; 95%CI, 0.68-1.74) compared with conventional DAPT. These findings suggest that a potent P2Y12 inhibitor-based SAPT following a short DAPT course (1-3 months) may represent a preferable treatment option, which is associated with similar ischemic, but lower bleeding risk, for patients undergoing PCI with newer-generation DES compared to standard conventional 12 months DAPT.

The question of whether SAPT using a potent oral P2Y12 inhibitor (ticagrelor or prasugrel) without aspirin (aspirin-free strategy) after primary PCI with a newest-generation thin-strut polymer-free drug-eluting stent is safe and effective compared to a conventional guideline-recommended 6- to 12-month DAPT course among patients with STEMI remains uncertain.

ELIGIBILITY:
Inclusion criteria

* Age ≥18 years.
* Subjects who have received DAPT consisting of aspirin and any of the commercially available P2Y12 receptor inhibitors (ticagrelor, prasugrel, or clopidogrel) at the time of STEMI diagnosis, or at the very latest at the time of primary PCI.
* Subjects with ≥1 acute infarct artery target vessel with ≥1 coronary artery stenosis in a native coronary artery with diameter from 2.25 to 4.0 mm who underwent successful primary PCI, defined as primary PCI with ≥1 Abluminus NP polymer-free sirolimus-based nanocarrier eluting stent (Concept Medical Inc., India) implantation, and final residual stenosis <30% by visual estimation or 20% by quantitative coronary angiography (QCA) [38].
* Subject willing to participate and able to understand, read and sign the informed consent form.

Exclusion criteria:

* Known allergy or intolerance to aspirin, ticagrelor, prasugrel, or sirolimus.
* Inability to adhere to DAPT for at least 6 months.
* Patient already on DAPT at index presentation due to recent PCI for chronic coronary syndrome (<6 months) or ACS (<12 months).
* Patient on chronic oral anticoagulation at index presentation.
* Patient with mechanical complication of STEMI.
* Patient with STEMI due to stent thrombosis.
* Planned non-cardiac surgery that cannot be postponed for at least 6 months.
* Participation or planned participation in another interventional clinical trial.
* Life expectancy <1 years.
* Pregnancy.
* Unwillingness or inability (e.g. physical or cognitive) to comply with study procedure, medication adherence and schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of major adverse cardiac and cerebrovascular events (MACCE) | 12 months
  Composite of all-cause death, non-fatal myocardial re-infarction, non-fatal stroke, urgent target vessel revascularization (PCI, or CABG), or Academic Research Consortium (ARC) definite/probable stent thrombosis
Rate of BARC class 3 or 5 major bleeding | 12 months
  Bleeding Academic Research Consortium (BARC) criteria

SECONDARY OUTCOMES:
Rate of any death | 12 months
  All-cause and cardiac death
Rate of any non-fatal myocardial re-infarction | 12 months
  Target vessel, non-target vessel, clinically indicated, non-clinically indicated
Rate of any revascularization | 12 months
  PCI or CABG, target lesion, non-target lesion, target vessel, non-target vessel, clinically indicated, non-clinically indicated
Rate of patient-oriented cardiac outcome (POCE) | 12 months
  Composite of all-cause death, any non-fatal myocardial re-infarction, or any revascularization
Rate of target lesion failure (TLF) | 12 months
  Composite of cardiac death, target vessel myocardial re-infarction, and clinically indicated target lesion revascularization
Rate of target vessel failure (TVF) | 12 months
  Cardiac death, target vessel myocardial re-infarction, and clinically indicated target vessel revascularization
Rate of fefinite or probable stent thrombosis | 12 months
  Academic Research Consortium (ARC) criteria
Rate of definite stent thrombosis | 12 months
  Academic Research Consortium (ARC) criteria
Rate of BARC ≥2 major bleeding | 12 months
  Bleeding Academic Research Consortium (BARC) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Iglesias, MD, Principal Investigator — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - Geneva University Hospitals, Geneva, Canton of Geneva
  - Zurich University Hospital, Zurich